CLINICAL TRIAL: NCT05515731
Title: Platelet Rich Plasma as a Treatment For Resistant Corneal Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alaa Gamal (Network)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, Alaa Gamal, Al-Azhar University, Egyptian Biomedical Research Network
Organization: Egyptian Biomedical Research Network (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38983
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Cornea Ulcer
MeSH Terms: conditions — Corneal Ulcer | interventions — Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous platelet-rich plasma eye drops (Experimental): Autologous platelet-rich plasma eye drops are derived from treatment of patients plasma using special process.
  Interventions: Biological: Autologous platelet-rich plasma (PRP) eye drops

INTERVENTIONS:
Biological: Autologous platelet-rich plasma (PRP) eye drops — Autologous platelet-rich plasma (PRP) eye drops are used as a sole or adjunctive therapy in many ophthalmological conditions including dry eye, macular holes, retinitis pigmentosa and perforated corneal ulcers. Actions of PRP in these conditions are attributed to the plethora of growth and healing factors concentrated in different PRP preparations.

SUMMARY:
This prospective study involved 14 patients aged > 18 years with RCUs not responding to conventional treatment. All patients were treated with E-PRP drops (one drop), preservative-free artificial tears, antibiotic eye drop four times daily and systemic vitamin A once daily for one month. All patients were examined at 1, 2, 4, 6 and 8 weeks after the treatment initiation. In each visit, the following parameters were assessed: best corrected visual acuity (BCVA), anterior segment, corneal healing, condition of the conjunctiva, presence of abnormal discharge and symptoms reported.

DETAILED DESCRIPTION:
The present prospective study involved 14 patients aged > 18 years with RCUs not responding to conventional treatment. All patients were treated with E-PRP drops (one drop), preservative-free artificial tears, antibiotic eye drop four times daily and systemic vitamin A once daily for one month. All patients were examined at 1, 2, 4, 6 and 8 weeks after the treatment initiation. In each visit, the following parameters were assessed: best corrected visual acuity (BCVA), anterior segment, corneal healing, condition of the conjunctiva, presence of abnormal discharge and symptoms reported.

ELIGIBILITY:
Inclusion Criteria:

* Resistant corneal ulcers

Exclusion Criteria:

* history of topical anesthetic abuse, diagnosed with corneal dystrophies, history of neurotrophic corneal ulcers or chemical burn ulcer. Other exclusion criteria were pregnancy of systemic diseases or therapies affecting platelets count e.g. aspirin.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain scale | 8 weeks
  Corneal pain as felt by the patient according to visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gomaa, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar University, Cairo, Egypt